CLINICAL TRIAL: NCT04333498
Title: Use of ARV Drug Levels in Dried Blood Spots to Assess and Manage ART Adherence in South Africa
Brief Title: Use of Antiretroviral (ARV) Drug Levels in Dried Blood Spots (DBS) to Assess and Manage ART Adherence in South Africa
Acronym: ADD-ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Research Foundation for Mental Hygiene, Inc. (Other); Desmond Tutu HIV Foundation (Other); University of Cape Town (Other); University of Colorado, Denver (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Robert Remien, Research Scientist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 7213; R01AI122300 (NIH)
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: Therapeutic Adherence and Compliance
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receiving Feedback From DBS (Experimental): This arm of participants will receive monthly feedback from medical providers on their adherence measured through DBS.
  Interventions: Behavioral: Feedback on DBS Concentrations

INTERVENTIONS:
Behavioral: Feedback on DBS Concentrations — The study team will examine the feasibility and acceptability of a feedback system based on DBS concentration amounts.

SUMMARY:
This is a prospective, pilot study of HIV-positive individuals who have been on tenofovir-containing antiretroviral therapy for at least 4 months. The overall goal of this research is to determine the feasibility of giving patients and their providers monthly feedback about Tenofovir-Diphosphate (TFV-DP) drug levels and to examine patient and provider behaviors in response to receiving this information. This study will build upon the Aim 1 observational study and the subsequent patient and providerFeedback Development Workgroups (FDWs).

DETAILED DESCRIPTION:
This is a prospective, pilot study of HIV-positive individuals who have been on tenofovir-containing antiretroviral therapy for at least 4 months. The overall goal of this research is to determine the feasibility of giving patients and their providers monthly feedback about Tenofovir-Diphosphate (TFV-DP) drug levels and to examine patient and provider behaviors in response to receiving this information. This study will build upon the Aim 1 observational study and the subsequent patient and provider Feedback Development Workgroups (FDWs).

The study team will consent a sample (N=60) of HIV-positive patients for monthly assessments, including blood specimen collections to assess TFV-DP drug levels. Participants enrolled in this prospective, pilot study will be randomized to either the intervention arm in which they will receive monthly feedback on their TFV-DP drug levels (Feedback Group; N=30) or the control arm in which they will receive no feedback on TFV-DP drug levels (No Feedback Group; N=30).

The study will take place at the Gugulethu Research Offices (GRO) of the Desmond Tutu HIV Foundation (DTHF) in Gugulethu, 15km outside Cape Town, South Africa (SA). Study participants will be recruited from patients attending one of four public-sector ART clinics in the Klipfontein Health District, Western Cape, including (1) Hannan Crusaid Treatment Centre, (2) Nyanga Clinic, (3) Gugulethu Clinic (NY1), and (4) Vuyani Clinic.

Enrollment will occur over 3-4 months, during which study staff will recruit an average of 15-20 participants per month, for a total of 60 participants. Participants will remain in the study for 5 months, attending a baseline and 4 subsequent monthly study visits. At each monthly visit, study staff will obtain venous blood samples for dried blood spots (DBS) which will measure TFV-DP levels and a viral load (VL) assay. ART adherence will also be assessed through the Wise Pill electronic monitoring device (EMD) a medication dispenser that sends an electronic medication event record to the Wisepill server when medication is taken and monthly self-reported medication adherence. Socio-demographic characteristics, medical history, mental health, substance use, and other contextual factors will be assessed at baseline and at the final study visit. In addition, at each visit, participants randomized to the intervention arm will receive feedback on their previous month's TFV-DP drug levels. Clinic providers will also receive TFV-DP drug level results for the participants in the intervention arm.

For both intervention and control groups, the study will monitor any changes to ART adherence behavior on the part of patients and providers. Potential changes will be monitored by reviewing participants' clinic charts to determine if any actions were made to the medical or adherence management of patients since the previous visit (e.g., additional VL requests beyond those prescribed for a stable patient, referral for intensive counselor-based or group adherence counseling, outreach by Health Care Workers (HCWs) for adherence monitoring and support, additional doctor-requested patient appointments). The study will also conduct Exit Interviews with participants and hold Provider Focus Group Discussions (FGD) to further understand whether (and if so, how) TFV-DP drug level feedback influenced medication adherence and patient management.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* HIV-positive
* Initiated ARV's containing tenofovir 4 or more months ago
* Speaks English or Xhosa
* Willing to attend 5 study visits approximately one month apart
* Willing to allow the study team to contact his/her HIV care provider about his/her monthly TFV-diphosphate (TFV-DP) drug level
* Willing to use Wise Pill to dispense ARVs for 4 months
* Willing to receive text/short message service (SMS) and/or phone call reminders to charge the Wise Pill
* Willing to allow the study team access to their medical chart/clinic folder

Exclusion Criteria:

* Unable to provide informed consent
* Unwilling to participate in study procedures
* Unwilling to allow the study team to contact his/her HIV care provider about his/her monthly TFV-DP drug level
* Any condition that, in the opinion of the principal investigator would make participation in the study unsafe, complicated interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Remien, Ph.D, Principal Investigator — NY State Psychiatric Institute: Columbia University Department of Psychiatry, College of Physicians and Surgeons; Catherine Orrell, Ph.D MBChB, Principal Investigator — Desmond Tutu HIV Centre/Foundation: University of Cape Town
Locations (2):
- 1051 Riverside Drive, New York, New York, United States
- Gugulethu Clinic, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 people with HIV (PWH) were recruited from an ART clinic in Cape Town. Recruitment commenced in 09/2020 and ended 02/2021.
Pre-assignment Details: No pre-assignment details to note, all participants were randomized on the day they were enrolled.
Groups:
- Receiving Feedback From TFV-DP Drug Levels Through DBS: This arm of participants will receive monthly feedback from research staff on their ART adherence measured through TFV-DP levels in dried blood spots (DBS). Adherence change in this group will later be measured through TFV-DP levels, Wisepill use, Viral Load, and self-report.
- No Feedback: This arm of participants will not receive monthly feedback through TFV-DP levels in DBS. This group is receiving standard of care (control).
Period: Overall Study
Arm/Group | Receiving Feedback From TFV-DP Drug Levels Through DBS | No Feedback
Started | 30 | 30
Completed | 29 | 29
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Receiving Feedback From TFV-DP Drug Levels Through DBS: This arm of participants will receive monthly feedback from medical providers on their adherence measured through DBS.
- No Feedback: This arm of participants will not receive monthly feedback through TFV-DP levels in DBS.
- Total: Total of all reporting groups
Arm/Group | Receiving Feedback From TFV-DP Drug Levels Through DBS | No Feedback | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [31 to 45] | 41 [32 to 47] | 39 [31 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 30 | 60
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 30 | 30 | 60
Hematocrit [Median (Inter-Quartile Range); unit: % of red blood cells] | 33 [31 to 35] | 32 [30 to 35] | 32 [30 to 35]
Months on ART [Median (Inter-Quartile Range); unit: Months] | 68 [45 to 128] | 52 [47 to 99] | 56 [47 to 108]
Baseline TFV-DP Result [Mean (Standard Deviation); unit: fmol/punch] | 1163 (856) | 1011 (433) | 1087 (677)

OUTCOME MEASURES:

1. Primary Outcome: TFV-diphosphate (TFV-DP) Drug Level
Description: Tenofovir diphosphate (TFV-DP) in dried blood spots (DBS) is used as a biomarker of antiretroviral therapy (ART) adherence. Recent treatment studies have shown that TFV-DP predicts future viremia in persons with HIV (PWH). Whole blood for DBS was collected at each study visit by venipuncture. To prepare the DBS, 25 mcl of whole blood were spotted five times onto a Whatman 903 ProteinSaver card and dried for a minimum of 3hrs and up to overnight before being individually packaged in a plastic bag with dessicant and a humidity indicator.
Time Frame: 5 Months
Measure: Mean (Standard Deviation); unit: fentomole/punch
Arm/Group | Receiving Feedback From TFV-DP Drug Levels Through DBS | No Feedback
Number analyzed (Participants) | 30 | 30
fentomole/punch | 1377.82 (846.45) | 1156.79 (653.99)
Statistical Analysis 1: Comparison: Receiving Feedback From TFV-DP Drug Levels Through DBS vs No Feedback; Test type: Other; p = .014, t-test, 2 sided; Mean Difference (Net) = -221.03, 95% CI 2-sided [-396.33 to -45.73]

2. Primary Outcome: Viral Load (VL) Assay
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: copies/ml
Arm/Group | Receiving Feedback From TFV-DP Drug Levels Through DBS | No Feedback
Number analyzed (Participants) | 30 | 30
copies/ml | 67.07 (622.12) | 1170.17 (8450.75)
Statistical Analysis 1: Comparison: Receiving Feedback From TFV-DP Drug Levels Through DBS vs No Feedback; Test type: Other; p = 0.122, t-test, 2 sided; Mean Difference (Net) = 1103.96, 95% CI 2-sided [-296.532 to 2502.722]

3. Primary Outcome: Electronic Adherence (EA) Percentages
Description: The number of days recorded as intake on electronic medical device (EMD) divided by days on study
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: Percentage of days recorded as intake
Arm/Group | Receiving Feedback From TFV-DP Drug Levels Through DBS | No Feedback
Number analyzed (Participants) | 30 | 30
Percentage of days recorded as intake | 81 (21) | 79 (22)
Statistical Analysis 1: Comparison: Receiving Feedback From TFV-DP Drug Levels Through DBS vs No Feedback; Adherence percentage; Test type: Other; p = .218, t-test, 2 sided; Mean Difference (Net) = -2.61, 95% CI 2-sided [-8.614 to 3.391]
Statistical Analysis 2: Comparison: Receiving Feedback From TFV-DP Drug Levels Through DBS vs No Feedback; Test type: Other — Linear regression with generalized estimating equations (GEE); p = 0.272, Regression, Linear; Slope = 0.046, 95% CI 2-sided [-0.036 to 0.128]

ADVERSE EVENTS:
Time Frame: 5 months (1st Baseline Visit + 4 subsequent study visits)
Arm/Group | Receiving Feedback From TFV-DP Drug Levels Through DBS | No Feedback
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT04333498/Prot_SAP_000.pdf